CLINICAL TRIAL: NCT05411510
Title: Evaluation of Bone Height Gain Following Trans-crestal Sinus Floor Elevation Using the Densifying Bur in Comparison to The Conventional Osteotome In Patients With Atrophic Posterior Maxillae: A Randomized Controlled Clinical Trial
Brief Title: Evaluation of Bone Height Gain Following Trans-crestal Sinus Floor Elevation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ahmed Mohamed Said Rozeik (Other)
Responsible Party: Sponsor-Investigator, Ahmed Mohamed Said Rozeik, Priniciple investigator, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022
Record Dates: First submitted 2022-05-20; First posted 2022-06-09 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Maxillary Sinus Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Densah bur (Experimental): According to the protocol for densah burs. The direction was reversed and the cutting speed was raised to 1200 rpm after the initial perforation close to the sinus floor. After that, two densifying burs were used in succession to elevate the sinus membrane by 2 mm and prepare the implant hole to the desired implant size.
  Interventions: Procedure: Densah bur
- Ostetome (Active Comparator): Flat end osteotome of appropriate size will be introduced through the osteotomy to infracture the floor of the sinus by light malleting.
  Interventions: Procedure: Densah bur

INTERVENTIONS:
Procedure: Densah bur — Surgical treatment
  Other Names: Densifying bur

SUMMARY:
Missing teeth usually result in functional and cosmetic deficits. Traditionally, they have been restored with dentures or fixed bridges. However, dental implants represent an excellent alternative which rely on the maintenance of a direct structural and functional connection between living bone and implant surface, which is termed osseointergration . When sufficient bone is available in maxilla, implant rehabilitation has shown high success rates of 84-92 %. Atrophy of the alveolar crest and pneumatization of the maxillary sinus limits the quality and quantity of residual bone, therefore complicating the placement of implants in the posterior maxillary area.

DETAILED DESCRIPTION:
Among the techniques used to overcome low vertical bone height in the maxilla is maxillary sinus floor augmentation. It can be performed either through a lateral window, or via a crestal access. Many long term studies and systematic reviews have showed that osteotome mediated sinus floor elevation (OSFE) technique is a highly predictable method for rehabilitation of patients with atrophied posterior maxilla with survival rates ranging from 92 % to 100 %. However, endoscopic studies have demonstrated the risk of membrane perforation while performing transalveolar sinus floor elevation. Moreover, the Summers technique can cause some complications as headache and paroxysmal positional vertigo. Additionally, the activity of osteotomes during the application of malleting pressure is difficult to control, resulting in unwanted instrument and/or graft penetration into the sinus cavity, potentially causing membrane penetration.

However, Huwais invented a new technology termed osseodensification for enhancing implant primary stability in 2015. This technology is performed with the use of specially developed drill bits (Densah burs) that combine the benefits of osteotomes with tactile control during the expansion. They have four or more lands with a negative rake angle, which prevents the bur's edges from cutting the bone and so compacts it smoothly. These drills have a tapered shank and a cutting chisel edge. They can thus go deeper into the osteotomy site, while the drill's gradually increasing diameter aids in the site's gradual enlargement. Drills are utilized to enter into the bone in a clockwise rotation (Cutting mode) until the appropriate depth of the osteotomy is reached. Afterwards, counterclockwise rotations (Densifying mode) generate a robust and dense layer of bone tissue along the osteotomy's walls and base. Through controlled deformation, this procedure burnishes bone along the inner layer of the osteotomy site. The goal is to construct a condensed layer of autografted bone along the implant's periphery and apex. This would improve the bone-implant contact, hence increasing insertion torque values and, as a result, implant primary stability.

ELIGIBILITY:
Inclusion Criteria:

* ● Patients having one missing upper posterior tooth with residual bone height beneath maxillary sinus from 5-8 mm.

  * A minimum of 6 mm residual bone width at site of implant placement.
  * The recipient site of the implant should be free from any pathological conditions.
  * No diagnosed bone disease or medication known to affect bone metabolism.
  * Patients who are cooperative, motivated and hygiene conscious.
  * Patients having adequate inter-occlusal space of 8-10 mm

Exclusion Criteria:

* ● Systemic conditions/diseases that contraindicate surgery.

  * Radiation therapy in the head and neck region or chemotherapy during the 12 months prior to surgery.
  * Patients who have any habits that might jeopardize the osseointegration process, such as current smokers.
  * Patients with parafunctional habits that produce overload on implant, such as bruxism and clenching.
  * Patients that have any pathology in the maxillary sinuses.

Ages: 23 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-08-20 (Estimated); Primary Completion 2023-02-20 (Estimated); Study Completion 2023-12-20 (Estimated)

PRIMARY OUTCOMES:
Bone gain height | 6 months
  It will be measured using Cone beam computed tomography (CBCT) in mm

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Cairo University, Cairo
  - Faculty of Dentistry, Cairo

IPD SHARING:
Plan to Share IPD: Undecided